CLINICAL TRIAL: NCT03306238
Title: Laparoscopic Entry Technique in Renal Surgery: a Randomised Controlled Trial Comparing Open (Hasson) Versus Closed (Veress) Techniques.
Brief Title: LAParoscopic Entry Technique in REnal Surgery
Acronym: LAPRES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Adelaide and Meath Hospital, incorporating The National Children's Hospital (Other)
Responsible Party: Principal Investigator, Arun Thomas, Principal investigator, The Adelaide and Meath Hospital, incorporating The National Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AMNCH-GU-2017-3
Record Dates: First submitted 2017-09-23; First posted 2017-10-11 (Actual); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Kidney Diseases
Keywords: laparoscopy/ key-hole; renal surgery; open/hasson; closed/veress
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Intervention Model Description: This is a randomised single blinded prospective trial comparing two similar groups directly to check for differnces in time to approach and complication rate
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The patient and the investigator will not be informed of the type of approach they had. These will be marked as A and B with only the care povide/surgeon being aware of the actual approach. The investigator of complications and assessor of the case outcomes will collect data without the knowledge of the group the patient belongs to. The surgeon or car eprovider cannot be masked in this case due to technical limitations but they will not contribute towards analysing the results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open/Hasson (Active Comparator): This group will undergo initial laparoscopic port insertion by the open or Hasson approach and then undergo the remaining laparoscopic surgery as usual
  Interventions: Procedure: Open approach to port insertion
- Closed/ Veress (Active Comparator): This group will undergo initial laparoscopic port insertion by the closed or Veress approach and then undergo the remaining laparoscopic surgery as usual
  Interventions: Procedure: Closed approach to port insertion

INTERVENTIONS:
Procedure: Open approach to port insertion — This involves the peritoneum being cut down, followed by the insertion of a blunt trocar under direct visualisation, gas insufflation, and insertion of the laparoscope
  Other Names: Hasson
  Arms: Open/Hasson
Procedure: Closed approach to port insertion — This involves the insertion of a Veress needle (a needle equipped with a spring-loaded obturator) into the peritoneal cavity, followed by gas insufflation (act of blowing) and insertion of a trocar (a sharp, pointed instrument with a cannula used to enter the body cavity).
  Other Names: Veress
  Arms: Closed/ Veress

SUMMARY:
This is a randomised controlled trial to evaluate safety and efficacy of two different port site entry techniques in laparoscopic renal surgery: open method (Hasson) and closed method (Veress). It will involve 300 adult patients undergoing elective laparoscopic renal surgery in Tallaght hospital under two Consultant urologists.

DETAILED DESCRIPTION:
Surgical specialties commonly using laparoscopic techniques like gynecology and general surgery have extensively compared the various available techniques of port insertion (1). There is very little known regarding the safest entry technique for the initial port in laparoscopic renal surgery. Results from other surgical specialties cannot simply be extrapolated to this type of laparoscopic surgery due to difference in entry site and patient position with renal surgery. Hence, this randomised controlled trial will be performed in a urological unit with two laparoscopic renal surgeons to compare two commonly used techniques of initial trocar insertion: the closed method and the open method.

Background Since its introduction in 1991 by Clayman, laparoscopic renal surgery has become very popular and is widely used for both benign and malignant renal operations such as radical, simple and partial nephrectomies, pyeloplasties, nephro-ureterectomies (2). The overall reported major and minor complication rate of laparoscopic renal surgery is 9.5% and 1.9% respectively (2). Initial entry by trocar insertion is the most hazardous part of the laparoscopic procedure. Opinion regarding the safest entry technique is divided. The two most commonly used techniques of port entry include open and closed (3). An open technique, as first described by Hasson, involves the peritoneum being cut down, followed by the insertion of a blunt trocar under direct visualisation, gas insufflation, and insertion of the laparoscope. One of the closed technique involves the insertion of a Veress needle (a needle equipped with a spring-loaded obturator) into the peritoneal cavity, followed by gas insufflation (act of blowing) and insertion of a trocar (a sharp, pointed instrument with a cannula used to enter the body cavity). Finally the laparoscope is passed through the trocar once the obturator is removed. Previous meta-analyses in laparoscopic surgery from gynaecological and general surgical operations have not been able to support one technique over the other due to insufficient evidence.to our knowledge (3), there are no randomised controlled trials comparing these two techniques in laparoscopic renal surgery. During laparoscopic renal surgery, the patient is placed in a lateral flank position with the table flexed. The initial port of entry can be either at the umbilicus or lateral to it. This position is unique to urological surgery and hence can have different implications to the initial trocar insertion technique.

The objective is to compare the open method (Hasson) and closed method (Veress) of laparoscopic port site entry in renal surgery

ELIGIBILITY:
Inclusion Criteria:

* • Able to undergo a general anaesthetic

  * At least 18 years old
  * Willing and able to give AN INFORMED CONSENT

Exclusion Criteria:

* patient refusal obese patients BMI >40mg/m2 previous laparotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Complications | 48 hours
  Minor and major complications assessed

SECONDARY OUTCOMES:
Time to insertion | 30 minutes
  Record time taken to perform both approaches

CONTACTS AND LOCATIONS:
Overall Officials: Arun Z Thomas, Principal Investigator — AMNCH, Tallaght hospital, Dublin 24
Locations (1):
- Adelaide and Meath hospital incorporating the NAtional Children's hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Angioli R, Terranova C, De Cicco Nardone C, Cafa EV, Damiani P, Portuesi R, Muzii L, Plotti F, Zullo MA, Panici PB. A comparison of three different entry techniques in gynecological laparoscopic surgery: a randomized prospective trial. Eur J Obstet Gynecol Reprod Biol. 2013 Dec;171(2):339-42. doi: 10.1016/j.ejogrb.2013.09.012. Epub 2013 Sep 23. PMID 24103531
- [Background] Pareek G, Hedican SP, Gee JR, Bruskewitz RC, Nakada SY. Meta-analysis of the complications of laparoscopic renal surgery: comparison of procedures and techniques. J Urol. 2006 Apr;175(4):1208-13. doi: 10.1016/S0022-5347(05)00639-7. PMID 16515961
- [Background] Ahmad G, O'Flynn H, Duffy JM, Phillips K, Watson A. Laparoscopic entry techniques. Cochrane Database Syst Rev. 2012 Feb 15;(2):CD006583. doi: 10.1002/14651858.CD006583.pub3. PMID 22336819